CLINICAL TRIAL: NCT02521844
Title: A Phase 1A/B Study to Evaluate the Safety and Tolerability of ETC-1922159 as a Single Agent and in Combination With Pembrolizumab in Advanced Solid Tumours
Brief Title: A Study to Evaluate the Safety and Tolerability of ETC-1922159 as a Single Agent and in Combination With Pembrolizumab in Advanced Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EDDC (Experimental Drug Development Centre), A*STAR Research Entities (Other Government)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3-002
Record Dates: First submitted 2015-07-27; First posted 2015-08-13 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: solid tumors; responsive to Wnt signalling regulation; RSPO fusions; Porcupine; PD-1; MSS; CRC; endometrial cancer; ovarian cancer
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms | interventions — ETC-159; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): ETC-1922159 + pembrolizumab
  Interventions: Drug: ETC-1922159; Drug: Pembrolizumab
- Dose Expansion (Experimental): ETC-1922159 as single agent until disease progression, then in combination with pembrolizumab at the recommended dose (RD) identified in the dose escalation segment
  Interventions: Drug: ETC-1922159; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ETC-1922159 — Oral administration
Drug: Pembrolizumab — IV administration

SUMMARY:
This is a Phase 1A/B study consisting of four parts.

1. Part A (completed) is a non-randomised, open-label, sequential evaluation of the safety, pharmacokinetics (PK), maximum tolerated dose (MTD), and recommended dose (RD) of ETC-1922159 in patients with advanced or metastatic, or unresectable solid malignancies, for whom no approved treatment option or standard of care is available. Dose escalation, with the goal of identifying the MTD and RD, is guided by an ordinal continual reassessment method (oCRM) model with a cohort size of one patient.
2. Part A extension (completed) is a non-randomised, non-comparative, open-label evaluation of the safety and tolerability of ETC-1922159 together with the bone protective treatment (denosumab) in patients with advanced or metastatic, or unresectable solid malignancies, for whom no approved treatment option or standard of care is available.
3. Part B dose escalation (completed) is a non-randomised, open-label, sequential evaluation of the MTD, RD, safety, PK, and PD (pharmacodynamics) of ETC 1922159 in combination with pembrolizumab in patients with advanced or metastatic, or unresectable solid malignancies, for whom no approved treatment option or standard of care is available.
4. Part B dose expansion will be a non-randomised, non-comparative, open-label study evaluation of the safety and tolerability of ETC-1922159 as a single agent until disease progression and then in combination with pembrolizumab at the RD identified in the Part B dose escalation segment, in patients with advanced or metastatic, or unresectable solid malignancies that are refractory, intolerant or not suitable for available treatment according to the treating physician.

It is anticipated that the study will take approximately 78 months to complete (36 months for Part A and Part A Extension, approximately 6 months for Part B dose escalation and approximately 36 months for Part B dose expansion).

ELIGIBILITY:
Inclusion Criteria (Part B):

* 18+ yrs (US), 21+ yrs (Singapore)
* Ability to give informed consent
* Histologically/cytologically confirmed advanced or metastatic tumors, that are unresectable solid malignancies, and that are are refractory, intolerant or not suitable to available treatment
* Objective and radiologically confirmed disease progression at screening
* Measurable disease by RECIST v1.1
* ECOG (Eastern Cooperative Oncology Group) 0-2
* Life expectancy ≥3 months
* Organ function:

  * Absolute neutrophil count ≥1.0×10^9/L
  * Platelets ≥100×10^9/L (w/o transfusions w/in 21 days)
  * Hemoglobin ≥9 g/dL
  * PT (prothrombin time) and PTT (partial thromboplastin time) w/in ≤1.5× ULN
  * International normalised ration (INR) ≤1.5× ULN Note: If the patient is on allowed anti-coagulants the INR should be in the therapeutic range
  * Total bilirubin ≤1.5× ULN
  * Transaminases (AST and/or alanine aminotransferase) ≤2.5× ULN (<5× ULN with liver metastases)
  * Creatinine clearance ≥60 mL/min
  * Total calcium (corrected for serum albumin) within normal limits

Note: Patients with grade 1 changes can be included as long as they are asymptomatic and can receive supplementation during the study.

* Magnesium ≥ lower limit of normal (LLN). Note: Patients with grade 1 changes can be included as long as they are asymptomatic and can receive supplementation during the study.
* Normal urinalysis

  * Patients must have a T-score greater than -1 to be eligible, however, patients with osteopenia (T-score of -1 to -2.5 at L/R total hip, L/R femoral neck or lumbar spine [L1-L4]) are eligible to participate and will receive calcium and vitamin D supplements during the study. Patients with osteoporosis (T-score of < -2.5) must be excluded.
  * Capable of swallowing study medication or has caregiver responsible for administering study drug
  * Negative serum pregnancy test
  * Dose Expansion - Group 1 and Group 2a only (patients with MSS or pMMR [microsatellite stable]-colorectal cancer [CRC]): Is refractory, intolerant or not suitable for treatment with fluoropyrimidine, oxaliplatin, or irinotecan.

Note: patients with advanced or metastatic appendiceal cancer refractory, intolerant to current standard of care, will be considered under the CRC cohort.

* Dose Expansion - Group 1 patients: MSS or pMMR-CRC with confirmed presence of at least one of the four different recurrent gene fusions involving RSPO2 or RSPO3 (Fusions A-D). Note: If adequate tissue samples are available as determined by the lab or pathologist, patients do not have to wait for the result before enrolment into Group 1 and Group 2a. Patients with indeterminate and/or unreported results may be enrolled into Group 2a, but can be retrospectively assigned to Group 1 once the patient has a confirmed RSPO gene fusion determined as described above.
* Dose Expansion - Group 2a patients: Has MSS or pMMR-CRC with confirmed absence of all four different recurrent gene fusions involving RSPO2 or RSPO3 (Fusions A-D).
* Dose Expansion - Groups 2b and 2c only (patients with MSS or pMMR-ovarian and MSS-endometrial cancer): Has advanced or metastatic disease for which further conventional therapy, e.g. platinum-based chemotherapy, is not suitable. Has MSS/pMMR tumours as determined by IHC (immunohistochemistry), PCR (polymerase chain reaction) or NGS (next generation sequencing).
* Dose expansion segment - Groups 2d only (MSS or pMMR cancers): Has advanced or metastatic disease for which further conventional therapy is not suitable according to the treating physician. Patients with MSS or pMMR solid tumours with molecular phenotypes potentially sensitive to upstream Wnt pathway inhibitors will be recruited.
* Dose Expansion: Pre-dose and post-dose tumour biopsies are mandatory unless tumour is inaccessible or deemed unsafe for procedure by principal investigator.
* Archival tumour tissue available (≥40 µm thickness with ≥20% tumour content; plus one 5-µm section for H&E stain:) for all patients that cannot provide a fresh tumour biopsy.

Exclusion Criteria (Part B):

* Male patient with sexual partner(s) of childbearing potential unwilling to use contraception. Sexually active male patients must use a condom during intercourse during the study and for 12 weeks after the end of treatment. Condom must also be used by vasectomised males.
* Female of childbearing potential, unless birth control is used during study and for 12 weeks after end of treatment.
* Pregnant or nursing (lactating) female.
* Dose Escalation: Current or anti-cancer therapy within 4 weeks pre-study or with Grade ≤1 side effects not resolved within 4 weeks pre-study.
* Dose Expansion segment: Has received previous treatment with pembrolizumab or immunotherapy treatment within 4 weeks (28 days) prior to starting the study drug is permitted

  * Dose Expansion (Groups 1, 2a, 2b and 2d): Immunotherapy within 4 weeks (28 days) prior to starting study.
  * Dose Expansion (Group 2c MSS endometrial cancer only): Immunotherapy either alone or in combination with lenvatinib within 4 weeks (28 days) prior starting study drug.
* Is receiving any concomitant anti-cancer therapy.
* Has used other investigational products within 4 weeks or 5 half-lives (whichever is longer) prior to first dose of study drug.
* Has evidence of other malignancy not in remission or history of other malignancy within last 3 yrs (exceptions: treated basal or skin squamous cell carcinoma or in situ cancer of cervix)
* Has central nervous system metastases, unless treated with surgery, whole brain radiation or stereotactic radiosurgery, and stable disease ≥8 weeks without steroid use for ≥4 weeks prior to first dose of study drug.
* Has received prior radiation therapy within 4 weeks, or limited field radiation within 2 weeks, prior to study drug, or with unresolved Grade ≤1 side effects.
* Has history of radiation to spine/pelvis bone or chemoradiation to pelvic organs in the last 6 months prior to starting study drug, or the side effects of such therapy have not resolved to Grade ≤1 (NOTE: Such patients can be enrolled as long as they do not have osteoporosis (for details of calculating T-score for eligibility see Inclusion Criterion 9). Patients should initiate concurrent bone protective treatment prophylaxis if any radiation therapy has been given in the last 2 years or they are at high risk of bone related AEs.
* Has had major surgical procedure within 4 weeks of starting study drug. Or patient has not fully recovered from all surgery-related complications to Grade ≤1.
* Has a history of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis.
* Has received bisphosphonate therapy for osteoporosis or symptomatic hypercalcaemia, or denosumab for osteoporosis prior to starting study drug.
* Has osteoporosis (T-score of < -2.5 at left or right total hip, left or right femoral neck, or lumbar spine [L1-L4] as determined by DEXA scan at Screening).
* Has a history of symptomatic vertebral fragility fractures or fragility fracture of hip, pelvis, wrist, or other location (fragility fracture - any fracture without trauma or as a result of a fall from ≤standing height).
* Has moderate (25%-40% decrease vertebral height) or severe (>40% decrease vertebral height) morphometric vertebral fractures.
* Has ß-CTX serum level >600 pg/mL in the morning after at least 10 hours of fasting at Screening. Note: If patients meet the exclusion criteria of ß-CTX serum level >600 pg/mL in the morning after at least 10 hours of fasting at screening, patient can begin their treatment with the bone protective treatment (denosumab with a starting dose of 120 mg, administered SC) as long as the patient has a ß-CTX serum level ≤1000 pg/mL.
* Has thyrotropin level less than lower limit of normal (LLN).
* Has 25-hydroxy vitamin D levels less than 25 mmol/L (10 ng/mL).
* Has bone metastases.
* Has a history of long QT or prolonged QTc (>460 ms).
* Is receiving, or has received thiazolidinedione peroxisome proliferator-activated receptor gamma agonist (e.g. Actos® [pioglitazone] and Avandia® [rosiglitazone]) w/in 4 wks prior to starting study drug.
* Has metabolic bone disease such as hyperparathyroidism, Paget's disease or osteomalacia.
* Has a known clinically significant bleeding disorder or coagulopathy.
* Is receiving or has received within 4 weeks prior to starting study drug, heparin, warfarin or similar anti-coagulants except for patients on low molecular weight heparin or Direct-Acting Oral Anticoagulants (DOACs: factor Xa or direct thrombin inhibitors) for treatment or prophylaxis.
* Has severe or unstable medical conditions such as heart failure, ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, ongoing cardiac arrhythmia requiring medication (Grade ≥2, by National Cancer Institute [NCI] CTCAE v. 4.03).
* Has a known history of human immunodeficiency virus (HIV) or active bacterial, viral or fungal infections.
* Has a history of gastric bypass surgery.
* Has received prior treatment with an inhibitor of the Wnt-B-catenin pathway.
* Is unwilling or unable to comply with the protocol.
* Cannot start treatment with the bone protective treatment with denosumab and/or zoledronic acid. Cannot start treatment with the bone protective treatment with denosumab SC, in patients requiring this treatment at the start of the study.
* Dose Expansion: Patient is unable to provide tumour tissue (from archival tissue or a fresh biopsy or tumour RNA).
* Has received prophylactic administration of hematopoietic colony stimulating factors within 4 weeks prior to starting study drug.
* Is receiving active treatment with an oral or IV glucocorticoid for ≥4 weeks at a daily dose equivalent to ≥10 mg of oral prednisone within the 12 weeks prior to starting the study drug.
* Has recent or current active infectious disease requiring systemic antibiotics or antifungal or antiviral treatment within 2 weeks prior to the start of the study drug. Subjects receiving prophylactic antibiotics (e.g. for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Has a serious non-healing wound.
* Has a history of vasculitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* Has received a live vaccine within 28 days prior to the start of study drug or anticipate that such live vaccine will be required during the study. Anti-SARS-CoV-2 live virus vaccines developed that utilised a replication-deficient simian adenoviral vector (ChAdOx1) should be avoided.

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ETC-1922159 when administered with pembrolizumab (Part B Dose Escalation) | For 2 cycles (42 days)
Recommended Dose (RD) of ETC-1922159 when administered with pembrolizumab (Part B Dose Escalation) | For 2 cycles (42 days)
Number of participants with adverse events (AEs) (Part B Dose Expansion) | From date of enrolment until end of treatment
Number of participants with adverse bone density imaging assessments via DEXA scan (Part B Dose Expansion) | From date of enrolment until end of treatment
Number of participants with abnormal 12-lead electrocardiogram (ECG) readings (Part B Dose Expansion) | From date of enrolment until end of treatment
Change in Eastern Cooperative Oncology Group performance status (Part B Dose Expansion) | From date of enrolment until end of treatment
Number of participants with abnormal clinical laboratory test results (Part B Dose Expansion) | From date of enrolment until end of treatment
Number of participants with abnormal vital sign measurements (Part B Dose Expansion) | From date of enrolment until end of treatment
Tolerability measured by monitoring of fatigue and gastrointestinal-related side effects and when applicable, immune-related side effects in patients (Part B Dose Expansion) | From date of enrolment until end of treatment

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) (Part B Dose Escalation) | From date of enrolment until end of treatment
Number of participants with adverse bone density imaging assessments via DEXA scan (Part B Dose Escalation) | From date of enrolment until end of treatment
Number of participants with abnormal 12-lead electrocardiogram (ECG) readings (Part B Dose Escalation) | From date of enrolment until end of treatment
Change in Eastern Cooperative Oncology Group performance status (Part B Dose Escalation) | From date of enrolment until end of treatment
Number of participants with abnormal clinical laboratory test results (Part B Dose Escalation) | From date of enrolment until end of treatment
Number of participants with abnormal vital sign measurements (Part B Dose Escalation) | From date of enrolment until end of treatment
Tolerability measured by monitoring of fatigue and gastrointestinal-related side effects and when applicable, immune-related side effects in patients (Part B Dose Escalation) | From date of enrolment until end of treatment
Clinical activity measured by RECIST (Response Evaluation Criteria in Solid Tumours) version 1.1 and iRECIST (Response Evaluation Criteria in Solid Tumours modified for immune-based therapeutics) (Part B Dose Expansion) | From date of enrolment until end of treatment
Clinical activity measured by RECIST (Response Evaluation Criteria in Solid Tumours) version 1.1 and iRECIST (Response Evaluation Criteria in Solid Tumours modified for immune-based therapeutics) (Part B Dose Escalation) | From date of enrolment until end of treatment
ETC-1922159 Maximum plasma concentration (Cmax) (Part B) | From date of enrolment until end of treatment
ETC-1922159 Area under the curve (AUC) (Part B) | From date of enrolment until end of treatment
Retrospective evaluation of plasma/serum concentration of pembrolizumab (Part B) | From date of enrolment to Cycle 2 for Dose Escalation and Cycle 1 of combination therapy for Dose Expansion
Retrospective evaluation of plasma/serum concentration of bone protective agents, if administered (Part B) | Before and after the first administration only

CONTACTS AND LOCATIONS:
Overall Officials: Venkateshan Srirangam Prativadibhayankara, Study Director — EDDC, Medical Director; Karuppan C Palaniappan, Study Director — PPD, Medical Director
Locations (11):
- United States (9):
  - University of Arizona Cancer Center, 3838 N. Campbell Avenue, RM 2111, Site 203, Tucson, Arizona
  - Chao Family Comprehensive Cancer Center,Stern Center for Cancer Clinical Trials and Research, 101 City Drive South, Site 209, Orange, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, 12648 East 17th Avenue; MSF 700, Site 202, Aurora, Colorado
  - University of Kansas Medical Center, 4350 Shawnee Mission Parkway, Suite 2310, MS 6004, Site 210, Fairway, Kansas
  - Washington University School of Medicine, Siteman Cancer Center, 4921 Parkview Place, Site 205, St Louis, Missouri
  - Duke University Medical Center, Duke Cancer Center, 20 Duke Medicine Circle, Site 206, Durham, North Carolina
  - Oregon Health and Science University-Knight Cancer Institute, 3485 S Bond Ave., Mail code 0C14CTSite 211, Portland, Oregon
  - Oregon Health and Science University, 3181 Southwest Sam Jackson Park Road, Mail Code Cr 9-4, Site 211, Portland, Oregon
  - Department of Investigational Cancer Therapeutics, 1400 Holcombe Blvd., Unit 455, Site 201, Houston, Texas
- Singapore (2):
  - National University Hospital, 1E Kent Ridge Road, NUHS Tower Block, Level 7, Site 101, Singapore
  - National Cancer Centre Singapore, 11 Hospital Drive, Site 102, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls